CLINICAL TRIAL: NCT00067665
Title: Hypertension in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Rajiv Agarwal, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (DK62030); R01DK062030 (NIH)
Record Dates: First submitted 2003-08-25; First posted 2003-08-27 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-01

CONDITIONS: Hypertension; Left Ventricular Hypertrophy
Keywords: hemodialysis
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — Ultrafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Control group of 50 patients where dry weight is not changed.
- 2 (Experimental): All patients participating in the trial require evaluation of dry-weight at each dialysis visit for evaluation. An initial weight loss of 0.1kg/10 kg body-weight will be prescribed per dialysis. If ultrafiltration is not tolerated based on muscle cramps, need for excessive saline or symptomatic hypotension, the intensity of ultrafiltration will be reduced by 50%. If ultrafiltration is still not tolerated, the weight loss will be further reduced by 50%. If the patient cannot tolerate at least 0.2 kg incremental weight loss per dialysis, the patient will be said to be at goal dry-weight. Thus, by this protocol, all patients must experience symptoms of volume depletion to be at dry weight.
  Interventions: Other: Ultrafiltration

INTERVENTIONS:
Other: Ultrafiltration — All patients participating in the trial require evaluation of dry-weight at each dialysis visit for evaluation. An initial weight loss of 0.1kg/10 kg body-weight will be prescribed per dialysis. If ultrafiltration is not tolerated based on muscle cramps, need for excessive saline or symptomatic hypotension, the intensity of ultrafiltration will be reduced by 50%. If ultrafiltration is still not tolerated, the weight loss will be further reduced by 50%. If the patient cannot tolerate at least 0.2 kg incremental weight loss per dialysis, the patient will be said to be at goal dry-weight. Thus, by this protocol, all patients must experience symptoms of volume depletion to be at dry weight.
  Arms: 2

SUMMARY:
How high blood pressure in hemodialysis patients should be diagnosed and treated using medications or without medications is the purpose of this study.

ELIGIBILITY:
- Adults with hypertension on hemodialysis Hypertensive, long-term (3 months or more) hemodialysis patients will be studied over a 6 hemodialysis baseline phase during which 44-hour interdialytic ambulatory BP will be performed and baseline symptoms collected. Patients with well-controlled hypertension, on anti-hypertensive therapy will have blood pressure medications withdrawn until they become hypertensive as assessed by 44-hour interdialytic ambulatory blood pressure recording. We will exclude patients who have had vascular event (stroke, myocardial infarction or limb ischemia requiring bypass) within previous six months, ambulatory BP >170 mm Hg systolic or >100 mm Hg diastolic, those who miss 2 or more hemodialysis treatments in the previous month, abuse street-drugs, require home oxygen, have symptomatic congestive heart failure or are morbidly obese (body mass index > 40 kg/m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2003-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome parameter will be systolic reduction in 44h-interdialytic ambulatory BP with ultrafiltration as compared to the control group by intention to treat analysis | 0, 4, 8 wks

SECONDARY OUTCOMES:
Per protocol analysis of primary outcome with 1. weight loss as the covariate. 2. baseline left-atrial size and weight loss as covariates.3. Others: (Description restricted by space limitation) | 0, 4, 8 wks

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Affiliated Dialysis Unit, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Agarwal R, Bouldin JM, Light RP, Garg A. Inferior vena cava diameter and left atrial diameter measure volume but not dry weight. Clin J Am Soc Nephrol. 2011 May;6(5):1066-72. doi: 10.2215/CJN.09321010. Epub 2011 Feb 17. PMID 21330484
- [Derived] Agarwal R, Light RP. Median intradialytic blood pressure can track changes evoked by probing dry-weight. Clin J Am Soc Nephrol. 2010 May;5(5):897-904. doi: 10.2215/CJN.08341109. Epub 2010 Feb 18. PMID 20167684
- [Derived] Sinha AD, Light RP, Agarwal R. Relative plasma volume monitoring during hemodialysis AIDS the assessment of dry weight. Hypertension. 2010 Feb;55(2):305-11. doi: 10.1161/HYPERTENSIONAHA.109.143974. Epub 2009 Dec 28. PMID 20038754
- [Derived] Agarwal R. Volume-associated ambulatory blood pressure patterns in hemodialysis patients. Hypertension. 2009 Aug;54(2):241-7. doi: 10.1161/HYPERTENSIONAHA.109.136366. Epub 2009 Jun 15. PMID 19528362
- [Derived] Agarwal R, Light RP. Chronobiology of arterial hypertension in hemodialysis patients: implications for home blood pressure monitoring. Am J Kidney Dis. 2009 Oct;54(4):693-701. doi: 10.1053/j.ajkd.2009.03.018. Epub 2009 Jun 10. PMID 19515473
- [Derived] Agarwal R, Alborzi P, Satyan S, Light RP. Dry-weight reduction in hypertensive hemodialysis patients (DRIP): a randomized, controlled trial. Hypertension. 2009 Mar;53(3):500-7. doi: 10.1161/HYPERTENSIONAHA.108.125674. Epub 2009 Jan 19. PMID 19153263